CLINICAL TRIAL: NCT01999361
Title: Myfortic® Monotherapy to Prevention of de Novo Allosensitization in Islet Transplant Recipients Following Complete Graft Loss
Brief Title: Prevention of de Novo Allosensitization in Islet Transplant Recipients Following Complete Graft Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rodolfo Alejandro (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20071058
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myfortic treatment (Experimental): Treatment with Myfortic
  Interventions: Drug: Myfortic

INTERVENTIONS:
Drug: Myfortic — treatment with myfortic
  Other Names: mycophenolic acid

SUMMARY:
This is a single-center, prospective, open label study in islet transplant recipients after complete islet graft rejection/loss, defined as stimulated c-peptide ≤0.3 ng/mL.

DETAILED DESCRIPTION:
After complete islet graft loss is determined, patient's maintenance immunosuppression (i.e. sirolimus and tacrolimus) will be discontinued and they will be placed on Myfortic® monotherapy for 2 years thereafter. After completion of two years of Myfortic® maintenance monotherapy, it will be weaned and subjects will be monitored over the subsequent twelve months, for the appearance of sensitization using panel reactive antibody (PRA) levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18-70 years of age.
2. Ability to provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study protocol.
4. Any subject currently prescribed immunosuppressive medications or discontinuation of immunosuppressive medications indicated as per current protocol of islet transplantation.
5. History of at least one islet transplant.
6. Stimulated C-peptide <0.3 ng/ml.

Exclusion Criteria:

1. Known history of untreated severe hyperlipidemia, obesity, or refractory hypertension
2. For female participants: Positive pregnancy test or presently breast-feeding.
3. History of active infection including hepatitis B, hepatitis C, HIV, or TB.
4. Any history of malignancy except for completely resected squamous or basal skin cell carcinoma.
5. Known active alcohol or substance abuse.
6. Severe co-existing history of cardiac disease, characterized by a history of any one of these conditions: recent myocardial infarction (within past 6 months), evidence of ischemia on functional cardiac exam within the last year, or left ventricular ejection fraction <30%.
7. History of persistent elevation of liver function tests. SGOT (AST), SGPT (ALT), alkaline phosphatase or total bilirubin, with values >1.5 times normal upper limits will exclude a patient.
8. Evidence of inter-current infection.
9. Active peptic ulcer disease
10. History on non-adherence to prescribed regimens including immunosuppression.
11. PRA ≥ 50% or evidence of significant sensitization to be determined at discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-01; Primary Completion 2027-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
allosensitization after complete islet graft loss | 3 years
  Allosensitization after complete islet graft loss after completion of two years of Myfortic® maintenance monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, MD, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rios P, Baidal D, Lemos J, Camhi SS, Infante M, Padilla N, Alvarez Gil AM, Fuenmayor V, Ambut J, Qasmi FA, Mantero AM, Cayetano SM, Ruiz P, Ricordi C, Alejandro R. Long-term Persistence of Allosensitization After Islet Allograft Failure. Transplantation. 2021 Nov 1;105(11):2490-2498. doi: 10.1097/TP.0000000000003635. PMID 33481552
- See also: Diabetes Research Institute clinical trials — https://diabetesresearch.org/dri-clinical-trials/